CLINICAL TRIAL: NCT00725062
Title: Phase I-II Dose Escalation Study of CD4+CD25+ Cells in Adult Patients Undergoing HLA-Identical Sibling Donor Peripheral Blood Progenitor Cell Transplantation
Brief Title: Donor T Cells in Treating Patients With High-Risk Hematologic Cancer Undergoing Donor Peripheral Blood Stem Cell Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004LS034; MT2004-03 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2008-07-29; First posted 2008-07-30 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: graft versus host disease; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients Receiving CD4+/CD25+ cells (Experimental): CD4+/CD25+ cells given intravenously over 15-60 minutes on Day -2 (prior to peripheral blood progenitor cell transplant)
  Interventions: Biological: CD4+CD25+ regulatory T cells; Procedure: allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: CD4+CD25+ regulatory T cells — Cohort 1 will receive 3 x 10^6 CD4+CD25+ cells/kg, Cohort 2 will receive 1 x 10^7 CD4+CD25+ cells/kg, Cohort 3 will receive 3 x 10^7 CD4+CD25 cells/kg
Procedure: allogeneic hematopoietic stem cell transplantation — Occurs on Day 0 of study - HLA-identical sibling donor peripheral blood progenitor cell (PBPC) transplantation
  Other Names: peripheral blood progenitor cell (PBPC) transplantation

SUMMARY:
RATIONALE: A donor peripheral stem cell transplant helps stop the growth of cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Once the donated stem cells begin working, the patient's immune system may see the remaining cancer cells as not belonging in the patient's body and destroy them. Giving an infusion of donor T cells may helps stop the patient's immune system from rejecting the donor's stem cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of donor T cells in treating patients with high-risk hematologic cancer who are undergoing donor peripheral blood stem cell transplant.

Note: Only Phase I portion of study was performed. Due to slow accrual, study was closed before Phase II portion of study.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose (MTD) of CD4+/CD25+ cells that can be safely administered to patients undergoing HLA-identical sibling donor Peripheral Blood Progenitor Cell (PBPC) transplantation.
* To determine whether CD4+ and CD25+ cells can be safely administered to patients with high-risk hematologic malignancies undergoing HLA-identical sibling donor PBPC transplantation.

Secondary

* To determine the incidence of grade II-IV acute graft-versus-host-disease (GVHD), chronic GVHD, relapse, and survival after administration of CD4+ and CD25+ regulatory T cells in these patients.

OUTLINE: This is a dose-escalation study of CD4+ and CD25+ donor regulatory T cells followed by a phase II study. All patients receive myeloablative preparative therapy and GVHD prophylaxis as per University of Minnesota protocol UMN-MT2001-02 or UMN-MT2001-10.

* First allogeneic peripheral blood progenitor cell (PBPC) infusion: Patients receive unmobilized, culture-expanded, CD4- and CD25-positive donor regulatory T cells IV over 15-60 minutes at the assigned dose on day -2.
* Second allogeneic PBPC infusion: Patients undergo matched-sibling donor PBPC transplantation IV on day 0.

Patients undergo blood sample collection prior to commencement of preparative therapy and then at day 100, 6 months, and 1 year after PBPC transplantation. Samples are analyzed for immune reconstitution by immunophenotyping and functional analyses.

After completion of study therapy, patients are followed for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a high-risk hematologic malignancy, including any of the following:

  * Acute lymphocytic leukemia
  * Acute myelocytic leukemia
  * Chronic myelogenous leukemia
  * Myelodysplastic syndrome
  * Non-Hodgkin lymphoma
  * Multiple myeloma
* Meet eligibility criteria and co-enrolled in one of the following University of Minnesota protocols:

  * MT2001-02 consisting of myeloablative prep (cyclophosphamide and total body irradiation) followed by HLA-identical sibling peripheral blood progenitor cells (PBPC) transplantation
  * MT2001-10 consisting of nonmyeloablative prep (cyclophosphamide, fludarabine and total body irradiation) followed by HLA-identical sibling PBPC transplantation
* Voluntarily written informed consent
* Must have an HLA-identical sibling donor available, meeting the following criteria:

  * 12 to 75 years of age, >40 kg body weight and in good health
  * Matched to recipient for HLA-A, B,DRB1 identical sibling match to recipient
  * Must be able and willing to have a separate apheresis collection performed on day -21 for the purposes of this study (in addition to the apheresis required for the transplant protocol)
  * Human immunodeficiency virus nucleic acid testing (HIV-NAT) negative, Human T-lymphotropic virus 1 (HTLV-1), HTLV-2 negative, hepatitic B and C negative

Exclusion Criteria:

* Not pregnant or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of CD4+CD25+ cells/kg (phase I) | Day 0 (48 hours post infusion)
Incidence of grade 3-5 infusional toxicity (phase II) | Day 0 (48 hours post infusion)

SECONDARY OUTCOMES:
Cumulative incidence of grade II-IV acute graft-versus-host-disease (GVHD) | Day 100 Post Infusion
Incidence of chronic graft-versus-host disease (GVHD) | Month 6 Post Infusion
Incidence of Relapse | Month 6 Post Infusion
Overall Survival | Day 100 and 1 Year Post Infusion
Disease-free survival | Day 100 and 1 Year Post Infusion

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L. MacMillan, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States